CLINICAL TRIAL: NCT07256912
Title: A Randomized, Active Controlled, Assessors-blind Trial to Establish Non-inferiority of Immunogenicity of a Single-dose of CERVAVAC® Quadrivalent HPV Vaccine Compared to the Gardasil® Quadrivalent Vaccine Among Girls and Boys Aged 9 to 14 Years and in Girls/Women Aged 15 to 20 Years in Zambia
Acronym: CervALONE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Responsible Party: Principal Investigator, Ravivarman Lakshmanasamy, Public Health Officer, International Agency for Research on Cancer
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CervALONE Trial
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Vaccine Effectiveness; HPV Vaccination; Single Dose; Immunogenicity
Keywords: HPV; VACCINE; SINGLE DOSE
MeSH Terms: interventions — Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Girls/women and boys vaccinated with single dose CERVAVAC vaccine (Experimental): CERVAVAC single dose vaccine will be administered - off label
  Interventions: Biological: HPV vaccine
- Girls/women and boys vaccinated with single dose Gardasil vaccine (Active Comparator)
  Interventions: Biological: HPV vaccine

INTERVENTIONS:
Biological: HPV vaccine — CERVAVAC single dose vaccine
  Other Names: CERVAVAC single dose
  Arms: Girls/women and boys vaccinated with single dose CERVAVAC vaccine
Biological: HPV vaccine — Gardasil-4 single dose
  Other Names: Gardasil-4 vaccine
  Arms: Girls/women and boys vaccinated with single dose Gardasil vaccine

SUMMARY:
The goal of this study is to compare the immune response of the single dose of the CERVAVAC vaccine with the single dose of Gardasil vaccine in girls/women aged 9 to 20 and boys aged 9 to 14 at 6 months, 12 months and 24 months post vaccination. The vaccine will be given randomly to the boys and girls/women in these age group and they will be followed up to check the immune status developed in them after vaccination. The status of immune response developed by the two differnet vaccines will be compared in these group of participants of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Girl/woman between 9 and 20 years of age and boy between the age of 9 and 14 years at the time of recruitment.
2. Participant willing to sign a written informed consent (for participants 18 years of age and above).
3. Parent (s) willing to provide written informed consent and participant is willing to sign written assent form for participation (for participants below 18 years of age at the time of eligibility assessment).
4. Participant or parent (s) willing to comply with all study requirements.
5. Participants who are determined by Medical History (MH), Physical Examination (PE) and clinical judgment of the Investigator to be eligible for inclusion in the study.

Exclusion Criteria:

1. Participants who are sexually active and missed their last menstrual period will have a urine pregnancy test and will be excluded if found pregnant.
2. Participant has a known history of prior vaccination with any HPV vaccine.
3. Participant known to be HIV positive (no routine HIV testing will be performed unless clinically indicated)
4. Participant currently enrolled in any other clinical studies of investigational products.
5. Participant with a current diagnosis or prior history of genital warts or treatment of genital warts.
6. Participant with a current diagnosis or prior history of cervical intraepithelial neoplasia (CIN) or cervical cancer.
7. Participant has a history of any allergic diseases or severe allergic reaction to any agent/vaccine product (e.g., swelling of the mouth and throat, difficulty in breathing, hypotension, or shock).
8. Participant has had an acute illness (moderate or severe) and/or fever (body temperature ≥ 38°C or ≥ 100.4 °F) at the time of vaccination or during the 72 hours prior to the vaccination.
9. Bleeding diathesis or uncontrolled condition associated with prolonged bleeding that would, in the opinion of the Investigator, contraindicate IM injection.
10. Participant has history of major congenital defects or illness that requires medical therapy, as determined by MH or clinical assessment.
11. Participant has had chronic administration (defined as more than 14 days) of high doses of corticosteroids (prednisone or equivalent at a dose of >0.5 mg/kg/day), cytotoxic agents or radiotherapy or immunoglobulins, immunosuppressants or other immune-modifying drugs in last 3 months or planned at any time during the study.
12. Participant has history of receiving a blood transfusion or other blood products in three months prior to screening.
13. Planned administration of a vaccine not foreseen by the study protocol within 14 days before and 14 days after any dose of study vaccine except TT given for emergency use and any vaccine mandated by government program.
14. Participant has history of any major pulmonary, cardiovascular, renal, neurological, metabolic, gastro-intestinal, hepato-biliary, hematological functional abnormality, mental or physical disability, blood dyscrasia or any condition which in the opinion of the Investigator might interfere with the evaluation of the study objectives.
15. Participant has history of any cancer, organ transplant or any other immune system disease.
16. Individuals who, in the opinion of the investigator, are unlikely to be compliant to all study procedures

Ages: 9 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1266 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Geometric mean Titre (GMT) of IgG antibodies against HPV 16 and 18 assessed from blood samples collected at 24 months and measured by M9ELISA on Meso-scale Discovery (MSD®) platform | 24 months

IPD SHARING:
Plan to Share IPD: Undecided